CLINICAL TRIAL: NCT04571593
Title: Digital Delivery of Yoga Nidra for Anxiety and Sleep: A Feasibility Study
Brief Title: Remote Yoga Nidra for Anxiety and Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Natural Medicine (Other)
Responsible Party: Principal Investigator, Erica Sharpe, Research Investigator, National University of Natural Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ESRB41320
Record Dates: First submitted 2020-09-17; First posted 2020-10-01 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Insomnia Due to Anxiety and Fear

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital Yoga Nidra (Experimental): Participants will voluntarily complete a ~30-minute remote Yoga Nidra practice, synchronously (through Zoom Wednesdays at 10 pm ET) or asynchronously (through YouTube, using the Zoom recording, any time they like).
  They may voluntarily repeat this practice as often as they like. Recordings are updated weekly, to reflect the ongoing Zoom class. Yoga Nidra scripts from Satyananda Saraswati's "Yoga Nidra" book (1976) are used for this class.
  Interventions: Behavioral: Yoga Nidra

INTERVENTIONS:
Behavioral: Yoga Nidra — The practice of Yoga Nidra, is a scripted and reproducible, guided meditation technique that promotes mental, emotional and physical relaxation while also facilitating the transition between waking and sleeping.

SUMMARY:
The goal of this application is to collect survey data indicating the effects of a digital Yoga Nidra practice on anxiety and sleep during COVID-19. We will explore effects on momentary anxiousness, as well as on sleep. Participants will be consented through REDCap during the Yoga Nidra class, then asked to complete an intake form, a sleep questionnaire (composed of questions from the Post Sleep Questionnaire (PSQ)) and a pre/post State Trait Anxiety (STAI) Index, surrounding the practice. Participants will receive an email the next morning, inquiring about their sleep (~2 min survey), and again the following week, the morning of the Yoga Nidra class, in order to remind them about the weekly class offering and also to collect sleep data for a night that did not include pre-bed Yoga Nidra. We will additionally report feasibility measures including enrollment, retention, qualitative feedback, and challenges of using the digital platform. Using this data, we will gain valuable feasibility data for implementation of this type of mind-body practice using digital platforms. We will also gain important data on the effects of this practice on anxiety and sleep.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Can understand a recording in English while resting comfortably

Exclusion Criteria: NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
Change in Momentary Anxiety | Pre-intervention and immediately after the intervention
  State Trait Anxiety (STAI-6) Short Form (scale 20 to 80, with higher scores indicating higher momentary anxiety)
Change in Sleep Quality | Baseline (pre-intervention), 1 day (morning after intervention), and 2-6 days later (survey sent each Tuesday, to capture a night without Yoga Nidra)
  Post Sleep Questionnaire (PSQ): six questions

SECONDARY OUTCOMES:
Incidence of Intervention-Emergent Challenges as assessed by a Feedback Survey | Post-intervention (survey sent at 16 weeks)
  Qualitative Feedback Survey (developed in-house)
Satisfaction as assessed by a Feedback Survey | Post-intervention (survey sent at 16-weeks)
  Qualitative Feedback Survey (developed in-house)

CONTACTS AND LOCATIONS:
Overall Officials: Erica M Sharpe, PhD, Principal Investigator — National University of Natural Medicine
Locations (1):
- National University of Natural Medicine, Helfgott Research Institute, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Protocol, analysis and consent are shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Available
Access Criteria: Uploaded to clinicaltrials.gov

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-04-13): https://cdn.clinicaltrials.gov/large-docs/93/NCT04571593/Prot_SAP_ICF_000.pdf